CLINICAL TRIAL: NCT06753279
Title: Clinical Significance of Leukocyte Cell Population Data in Patients with Myeloproliferative Neoplasms (MPNs)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ola Gamal Taha Hussein, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: leukocyte cell population MPNs
Record Dates: First submitted 2024-12-22; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Myeloproliferative Neoplasms (MPNs)
Keywords: leukocyte cell
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- cases: patients with MPNs according to the recent WHO classification
- control: normal healthy individual

SUMMARY:
Myeloproliferative neoplasms (MPNs) are a group of clonal hematopoietic disorders which categorized according to the World Health Organization (WHO) into Philadelphia Chromosome positive (Ph +ve) including chronic myeloid leukemia (CML) and Philadelphia Chromosome negative (Ph -ve) like essential thrombocythemia (ET), polycythaemia vera (PV), and primary myelofibrosis (PMF) .

the aim of the study is to Detection of leukocyte cell population data in patients with MPNs and Relation between leukocyte cell population and patients' clinical status.

DETAILED DESCRIPTION:
MPNs are characterized by sepsis, thrombosis, myelofibrosis and leukemic transformation as critical complications of the disease. Most recently, the MPNs have been described as "Inflammatory Diseases" because the chronic inflammation being identified as a key factor in the development and progression of the disease . It is characterized by persistent activation of immune cells, elevated leukocyte and platelet counts, release of various mediators, DNA and tissue damage . Consequently. when neutrophils are activated by different stimuli, they undergo degranulation and release neutrophil extracellular traps (NETs) and microparticles, leading to thrombosis in MPNs by blocking blood vessels . Monocyte and its distribution are also a simple marker of activation useful for early sepsis detection .

The leukocyte cell population data (CPD) are parameters used to provide quantitative information on the morphological and functional characteristics of leukocytes. CPD assessment involves measuring neutrophil and monocyte forward scatter (Z axis) for cell size and side scatter (X axis) for internal complexity. Additionally, fluorescence intensity (Y axis) for DNA/RNA content and cell population variability (dispersion width) can also be evaluated.

Therefore, assessing of these parameters in the context of sepsis and thrombosis as a complication of MPNs helps to understand how these conditions interact at the cellular level and provides insights into morphological changes and abnormal leukocyte distribution for early detection and management .

ELIGIBILITY:
Inclusion Criteria:

* Patients with MPNs according to the recent WHO classification.

Exclusion Criteria:

* Patients with other types of myeloid neoplasms and/or not fulfil the WHO criteria for MPNs diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: - Patients with MPNs according to the recent WHO classification.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
percentage of leukocyte cell in patients with MPNs | baseline
  Detection of leukocyte cell population data in patients with MPNs

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mishra S, Chhabra G, Padhi S, Mohapatra S, Panigrahi A, Sable MN, Das PK. Usefulness of Leucocyte Cell Population Data by Sysmex XN1000 Hematology Analyzer in Rapid Identification of Acute Leukemia. Indian J Hematol Blood Transfus. 2022 Jul;38(3):499-507. doi: 10.1007/s12288-021-01488-9. Epub 2021 Sep 28. PMID 35747581
- [Background] Camara JE, Wise SA, Hoofnagle AN, Williams EL, Carter GD, Jones J, Burdette CQ, Hahm G, Nalin F, Kuszak AJ, Merkel J, Durazo-Arvizu RA, Lukas P, Cavalier E, Popp C, Beckert C, Schultess J, Van Slooten G, Tourneur C, Pease C, Kaul R, Villarreal A, Ivison F, Fischer R, van den Ouweland JMW, Ho CS, Law EWK, Simard JN, Gonthier R, Holmquist B, Batista MC, Pham H, Bennett A, Meadows S, Cox L, Jansen E, Khan DA, Robyak K, Creer MH, Kilbane M, Twomey PJ, Freeman J, Parker N, Yuan J, Fitzgerald R, Mushtaq S, Clarke MW, Breen N, Simpson C, Sempos CT. Assessment of serum total 25-hydroxyvitamin D assay commutability of Standard Reference Materials and College of American Pathologists Accuracy-Based Vitamin D (ABVD) Scheme and Vitamin D External Quality Assessment Scheme (DEQAS) materials: Vitamin D Standardization Program (VDSP) Commutability Study 2. Anal Bioanal Chem. 2021 Aug;413(20):5067-5084. doi: 10.1007/s00216-021-03470-w. Epub 2021 Jun 28. PMID 34184102
- [Background] Hasselbalch HC. Chronic inflammation as a promotor of mutagenesis in essential thrombocythemia, polycythemia vera and myelofibrosis. A human inflammation model for cancer development? Leuk Res. 2013 Feb;37(2):214-20. doi: 10.1016/j.leukres.2012.10.020. Epub 2012 Nov 20. PMID 23174192